CLINICAL TRIAL: NCT00013195
Title: Nurse Counseling for Physical Activity in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NRM 95-022
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Disease; Exercise
Keywords: Telephone
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telephone Care

INTERVENTIONS:
Behavioral: Telephone Care

SUMMARY:
Many elderly primary care patients are at high risk for health complications and functional impairment due to low levels of physical activity. Previous trials of counseling of elderly patients in primary care clinics have not demonstrated lasting physical activity change and have not evaluated fitness changes associated with any increased activity.

DETAILED DESCRIPTION:
Background:

Many elderly primary care patients are at high risk for health complications and functional impairment due to low levels of physical activity. Previous trials of counseling of elderly patients in primary care clinics have not demonstrated lasting physical activity change and have not evaluated fitness changes associated with any increased activity.

Objectives:

The primary objective was to determine if nurse telephone counseling could assist 60 to 80 year old VA primary care patients to establish and maintain a regular walking program.

Methods:

In this randomized clinical trial, 60-80 year old patients were referred to a walking program by primary care providers. All participants received individualized counseling by the nurse and, over the next year, one of three follow-up interventions: 1) 20 calls initiated by the nurse; 2) ten calls initiated by the nurse and ten initiated by an automated telephone message delivery system; or 3) no follow-up calls. All kept walking diaries and mailed these in to a data collector blinded to intervention group. Follow-up research visits were scheduled at six and 12 months. Self-reported walking, the primary outcome measure, was assessed from the walking diaries and validated by reports of significant others and accelerometer data. Improvement in fitness was assessed at 12 months with a standardized six minute walking test. Tinetti mobility scores, body mass index, and body girths were also assessed. Several quality of life measures were also administered.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

60-80 year old patients referred to a walking program by a primary care provider.

Exclusion Criteria:

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Dubbert, PhD, Principal Investigator — G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS
Locations (1):
- G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jacksonport, Arkansas, United States

REFERENCES:
- [Result] Dubbert PM, Vander Weg MW, Kirchner KA, Shaw B. Evaluation of the 7-day physical activity recall in urban and rural men. Med Sci Sports Exerc. 2004 Sep;36(9):1646-54. doi: 10.1249/01.mss.0000139893.65189.f2. PMID 15354050
- [Result] Dubbert PM, Cooper KM, Kirchner KA, Meydrech EF, Bilbrew D. Effects of nurse counseling on walking for exercise in elderly primary care patients. J Gerontol A Biol Sci Med Sci. 2002 Nov;57(11):M733-40. doi: 10.1093/gerona/57.11.m733. PMID 12403802
- [Result] Dubbert PM, Meydrech EF, Kirchner KA, Cooper KM, Bilbrew DE. Encouraging elders to exercise. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2001 Jul 1; 18(7):39-59.
- [Result] Rhudy JL, Dubbert PM, Kirchner KA, Williams AE. Efficacy of a program to encourage walking in VA elderly primary care patients: the role of pain. Psychol Health Med. 2007 May;12(3):289-98. doi: 10.1080/13548500600986559. PMID 17510898
- [Result] Cooper TV, Resor MR, Stoever CJ, Dubbert PM. Physical activity and physical activity adherence in the elderly based on smoking status. Addict Behav. 2007 Oct;32(10):2268-73. doi: 10.1016/j.addbeh.2007.01.007. Epub 2007 Jan 11. PMID 17275199
- [Result] Cooper KM, Bilbrew D, Dubbert PM, Kerr K, Kirchner K. Health barriers to walking for exercise in elderly primary care. Geriatr Nurs. 2001 Sep-Oct;22(5):258-62. doi: 10.1067/mgn.2001.119470. PMID 11606904
- [Derived] Dubbert PM, Morey MC, Kirchner KA, Meydrech EF, Grothe K. Counseling for home-based walking and strength exercise in older primary care patients. Arch Intern Med. 2008 May 12;168(9):979-86. doi: 10.1001/archinte.168.9.979. PMID 18474762